CLINICAL TRIAL: NCT07373639
Title: A Long-term Follow-up Study in Patients With Hemoglobinopathy Who Received Autologous CD34+ Edited Hematopoietic Stem Cells
Brief Title: A Long-term Follow-up Study in Patients Who Received BEAM-101
Status: Recruiting | Type: Observational
Sponsor: Beam Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BTX-101-002
Record Dates: First submitted 2026-01-06; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Hemoglobinopathy; Sickle Cell Disease
MeSH Terms: conditions — Hemoglobinopathies; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BTX-101-002 Long-term Follow-up on Patients who received BEAM-101: All participants who received BEAM-101 in the BTX-AUT-001 trial will be asked to participate in this long-term follow-up study
  Interventions: Drug: Long-Term Follow-up Study of patients who received BEAM-101

INTERVENTIONS:
Drug: Long-Term Follow-up Study of patients who received BEAM-101 — This is a Long-Term Follow-up Study of patients who received a single dose of BEAM-101 administered by IV following myeloablative conditioning with busulfan

SUMMARY:
This is a Long-term Follow-up (LTFU) study in patients who received BEAM-101 in the parent study (Study BTX-AUT-001). Eligible patients who received BEAM-101 will be asked to participate in this LTFU study prior to completing Study BTX-AUT-001. Patients who enter into this study will be followed for 13 years (a total of 15 years after receiving BEAM-101).

DETAILED DESCRIPTION:
Patients who were treated with BEAM-101 in Study BTX-AUT-001 will be asked to sign an informed consent form (ICF) to enter this LTFU study (during the EOS/Month 24 visit for BTX-AUT-001). Patients in this study will have periodic safety and efficacy assessments per the schedule of assessments (SoA). Visits will occur annually through Year 5 following BEAM-101 administration and then every 3 years through Year 11, with a final visit at Year 15. Virtual/phone call check-in visits will occur every 6 months through Year 5 and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Have received BEAM-101 in Study BTX-AUT-001 and are in the process of completing that study's end-of-study (EOS) visit.
2. Provide signed, written informed consent according to local institutional review board (IRB)/independent ethics committee (IEC) and institutional requirements.

Exclusion Criteria:

* There are no exclusion criteria for this study.

Ages: 14 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of participants enrolled at sites from the parent study (BTX-AUT-001) who meet the criteria for long-term follow-up
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2043-02-12 (Estimated); Study Completion 2043-02-12 (Estimated)

PRIMARY OUTCOMES:
Long-Term Safety Monitoring and Mortality Assessment | Up to 13 years
  Monitor all BEAM-101-related AEs and SAEs through Year 15 post-IMP administration, all SAEs regardless of relatedness through Year 5, new malignancies, new or worsening bone marrow-related hematologic disorders, and all-cause mortality.

SECONDARY OUTCOMES:
Proportion of patients without severe VOCs overtime | Through year 15
Duration of being severe VOC-free | Through year 15
Frequency of RBC transfusions over time | Through year 15
Proportion (%) of patients requiring treatment for SCD related complications | Through year 15
Total Hemoglobin (Hb) Concentration (g/dL) over time | Through year 15
Total Fetal Hemoglobin (HbF) Concentration (%) over time | Through year 15
Total Sickle Hemoglobin (HbS) Concentration (%) | Through year 15
Change from baseline in indirect bilirubin (mg/dL) overtime | Up to year 5
Change from baseline in haptoglobin (mg/dL) over time | Up to year 5
Change from baseline in reticulocyte (%) count over time | Up to year 5

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Children's Healthcare of Atlanta - Aflac Cancer and Blood Disorders Center- Egleston, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Henry Ford Cancer Center, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - University Hospitals Clevland Medical Center, Cleveland, Ohio
  - The Clevland Clinic Foundation, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No